CLINICAL TRIAL: NCT03973450
Title: Epidemiology of Pituitary Tumours: Prevalence of Associated Endocrine and Non-endocrine Tumours and Potential Implications in the Management and Follow-up of Patients"
Brief Title: Epidemiology of Pituitary Tumours: Prevalence of Associated Neoplasia
Acronym: EpidemioPIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Marie-Lise Jaffrain-Rea, MD, Associate Professor of Endocrinology, Neuromed IRCCS
Other Study IDs: Neuroendo-1
Record Dates: First submitted 2019-05-25; First posted 2019-06-04 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Pituitary Tumor; Endocrine Neoplasia; Hyperparathyroidism; Solid Tumor; Familial Tumor Syndrome
MeSH Terms: conditions — Pituitary Neoplasms; Endocrine Gland Neoplasms; Hyperparathyroidism; Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pituitary tumours: Patients affected by pituitary tumours and followed-up at the Neuroendocrinology Unit over a 5 yrs period (2014-2018)
  Interventions: Other: Registration of familial forms and associated neoplasia

INTERVENTIONS:
Other: Registration of familial forms and associated neoplasia — Retrospective registration of associated endocrine and non-endocrine neoplasia and potential familial setting
  Other Names: Genetic counselling where appropriate

SUMMARY:
The study aims to update current knowledge about the epidemiology of pituitary tumours (PiT), based on the wide body of scientific literature on new familial and/or syndromic forms. Although inherited predisposition is increasingly recognized, its clinical relevance in unselected series of PiT patients has not been specifically addressed. In addition, it is likely that further recognition of peculiar associations between PiT and other endocrine and/or non-endocrine neoplasia will further increase the spectrum of syndromic forms. Since the identification of inherited forms of PiT may have significant clinical implications in terms of patients management and familial screening, we aim to collect any relevant information in order to estimate their prevalence in a large unselected series of PiT patients and provide new clues for a modern clinical approach to these patients.

DETAILED DESCRIPTION:
Recent epidemiological studies indicate that clinically relevant PiT have a prevalence around 1%. The Neuromed Scientific Institute for Research and Cure (IRCCS) is a third referral center for the diagnosis and treatment of patients with hypothalamic-pituitary disorders, and PiT represent the most frequent condition.

The best known syndromic of PiT is Multiple Endocrine Neoplasia type 1 (MEN1), others are rare conditions, such as MEN1-like syndromes, Carney complex, Mc Cune Albright syndrome, the pheochromocytoma/paraganglioma/Pit syndrome. Apparently isolated familial forms of PiT (FIPA) have also been well characterized in the last decade.The genetics of inherited PiT is involving a growing number of genes.At the moment, the most frequently reported gene abnormalities consist of inactivating mutations of the MEN1 and Aryl hydrocarbon receptor Interacting Protein (AIP) genes, which are mainly observed in syndromic and isolated familial forms of PiT, respectively.

On the other hand, patients affected by growth-hormone (GH)-secreting PiT (acromegaly/gigantism) have an increased risk of associated neoplasia, which has been mainly attributed to the growth-promoting effects of GH and/or Insulin-like Growth Factor 1(IGF1). However, a variety of neoplasia have been recently observed in patients with non-functioning PiT, whereas patients affected by prolactinoma - the most common PiT phenotype - have been poorly studied. Associations between PiT and a variety of neoplasia may represent new forms of systemic forms of PiT.

The aim of the study is to evaluate the prevalence of endocrine and non-endocrine neoplasia in a large series of PiTpatients and to identify potential familial and syndromic forms, including new forms of tumor associations, in order to provide new insights in the epidemiology and genetics of PiT and evaluate their clinical relevance in daily practice.

Eligible patients will receive a detailed informative form about the aim, methods and potential implications of the study. They will be included upon written informed consent and be re-assured that they may refuse to participate or withdraw from the study at any time, without any prejudice in their clinical management.

Data will be collected retrospectively in patients followed-up in the last 5 years, when an increased awareness of systemic conditions has lead, in the respect of good clinical practice, to a systematic registration of familiarity for PiT and/or for associated neoplasia. As clinically recommended, most patients have been screened at least once for primary hyperparathyroidism (pHPT), which is the most prevalent endocrine tumor in MEN1, and thyroid ultrasound, which is generally proposed as an extension of any endocrinological visit. Therefore, parathyroid and/or thyroid tumours should have been correctly identified in a large majority of patients. In contrast, except for systemic search for colonic polyps or tumours by coloscopy in acromegalic patients, and screening for breast and colon cancer performed by the patients in the setting of the Italian National Health System (NHS) programme since the age of 50 yr-old, no systematic search for additional tumours was performed and diagnoses were typically made by the general practitioner and other specialists.

Any relevant clinical, biological or imaging data about PiT and extrapituitary tumours will be collected for each patients.

All data will be collected anonymously in a dedicated Excel file.

Statistical analysis will be performed with using a commercially available software - JMP version 11.0 distributed by Statistical Analysis Systems (SAS) (USA). The first part of the report will be descriptive, report all endocrine and non-endocrine neoplasia and potential familiarity for PiT and/or any other associated neoplasia. Then, a comparison will be made between groups and subgroups of PiT patients defined according to the PiT phenotype (functioning and nonfunctioning PiT subgroups, tumour volume and invasiveness), as well as gender, age and the presence of a familial setting. Based on public reports of the Italian registry of cancer (AIRTUM), an attempt will be made to compare the prevalence of the most frequent neoplasia in PiT patients with the general population. Attention will be paid to recognize syndromic forms of PiT, including known syndromes and new forms of associations between PiT and any endocrine or non-endocrine neoplasia.

Genetic evaluation and counselling will be proposed in selected cases, based on evaluation of the clinical picture with the specialist in clinical genetics present in the study team. A specific additional consent will be necessary to proceed to the genetic step and DNA conservation for further studies where appropriate. Leukocyte DNA will be collected by blood sampling. Diagnostic genetic testing will be appropriately performed according to the clinical presentation. For unknown associations, this study is intended to be preliminary to further genetic studies aiming to identify new candidate genes.

ELIGIBILITY:
Inclusion Criteria:

* Any patient affected by a documented endocrine pituitary tumour (PiT)
* At least one evaluation during the study period (2014-2018)

Exclusion Criteria:

* Uncertain diagnosis of endocrine pituitary tumour
* Any adult patient declining to enter the study
* For the (few) patients aged less than 18 years, parents or legal tutors declining to include the patient in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We estimate that more than 500 patients followed at the Neuroendocrinology unit meet the eligibility criteria for the study period, and that a majority of them will accept to enter the study. Patients are affected prevalently by functional pituitary tumours (prolactinomas about 50%, followed by acromegaly about 20%, corticotroph tumours..), others have clinically non-functiong pituitary tumours (about 25%). The large majority of patients are adult (> 90 %).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hyperparathyroidism (HPT) | Up to 6 months
  measurement of plasma Parathormone (PTH) in % of upper limit of normal values (ULN)
Prevalence of hypercalcemia (hypercalcemic hyperparathyroidism) | Up to 6 months
  measurement of calcemia (mg/dl)
Search for secondary cause of hyperparathyroidism (1): vit D deficiency | Up to 6 months (where indicated)
  measurement of plasma 25(OH)D (ng/ml)
Search for secondary cause of hyperparathyroidism (2): renal failure | Up to 6 months
  measurement of plasma creatinine (mg/dl)
Prevalence of thyroid nodules | Up to 6 months
  Thyroid ultrasound
Prevalence of other endocrine and non-endocrine neoplasia (1) | Up to 6 months
  Report of any neoplasia before the diagnosis of PiT
Prevalence of other endocrine and non-endocrine neoplasia (2) | Up to 6 months
  Report of any neoplasia diagnosed during the follow-up of PiT
Familial setting (1) | Up to 6 months
  Report of any available information concerning familiarity for PiT
Familial setting (2) | up to 6 months
  Familiarity for any associated neoplasia

SECONDARY OUTCOMES:
Genetics (1) familial forms of PiT | up to 15 months
  AIP gene sequencing upon genetic counselling
Genetics (2) familial PiT and/or association with HPT | up to 15 months
  MEN1 sequencing upon genetic counselling
Genetics (3) any other clinical suspicion for MEN1 | up to 15 months
  MEN1 gene sequencing upon genetic counselling
Genetics (4) any other clinical suspicion of inherited neoplasia syndrome | up to 15 months
  genetic counselling for appropriate gene sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Lise Jaffrain-Rea, MD, Principal Investigator — Neuromed IRCCS, Pozzilli (IS), Italy
Locations (1):
- Neuromed, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daly AF, Rixhon M, Adam C, Dempegioti A, Tichomirowa MA, Beckers A. High prevalence of pituitary adenomas: a cross-sectional study in the province of Liege, Belgium. J Clin Endocrinol Metab. 2006 Dec;91(12):4769-75. doi: 10.1210/jc.2006-1668. Epub 2006 Sep 12. PMID 16968795
- [Background] Fernandez A, Karavitaki N, Wass JA. Prevalence of pituitary adenomas: a community-based, cross-sectional study in Banbury (Oxfordshire, UK). Clin Endocrinol (Oxf). 2010 Mar;72(3):377-82. doi: 10.1111/j.1365-2265.2009.03667.x. Epub 2009 Jul 24. PMID 19650784
- [Background] Caimari F, Korbonits M. Novel Genetic Causes of Pituitary Adenomas. Clin Cancer Res. 2016 Oct 15;22(20):5030-5042. doi: 10.1158/1078-0432.CCR-16-0452. PMID 27742789
- [Background] Corbetta S, Pizzocaro A, Peracchi M, Beck-Peccoz P, Faglia G, Spada A. Multiple endocrine neoplasia type 1 in patients with recognized pituitary tumours of different types. Clin Endocrinol (Oxf). 1997 Nov;47(5):507-12. doi: 10.1046/j.1365-2265.1997.3311122.x. PMID 9425388
- [Background] Alrezk R, Hannah-Shmouni F, Stratakis CA. MEN4 and CDKN1B mutations: the latest of the MEN syndromes. Endocr Relat Cancer. 2017 Oct;24(10):T195-T208. doi: 10.1530/ERC-17-0243. Epub 2017 Aug 19. PMID 28824003
- [Background] Thakker RV, Newey PJ, Walls GV, Bilezikian J, Dralle H, Ebeling PR, Melmed S, Sakurai A, Tonelli F, Brandi ML; Endocrine Society. Clinical practice guidelines for multiple endocrine neoplasia type 1 (MEN1). J Clin Endocrinol Metab. 2012 Sep;97(9):2990-3011. doi: 10.1210/jc.2012-1230. Epub 2012 Jun 20. PMID 22723327
- [Background] Olsson DS, Hammarstrand C, Bryngelsson IL, Nilsson AG, Andersson E, Johannsson G, Ragnarsson O. Incidence of malignant tumours in patients with a non-functioning pituitary adenoma. Endocr Relat Cancer. 2017 May;24(5):227-235. doi: 10.1530/ERC-16-0518. Epub 2017 Mar 8. PMID 28274953
- [Background] Terzolo M, Reimondo G, Berchialla P, Ferrante E, Malchiodi E, De Marinis L, Pivonello R, Grottoli S, Losa M, Cannavo S, Ferone D, Montini M, Bondanelli M, De Menis E, Martini C, Puxeddu E, Velardo A, Peri A, Faustini-Fustini M, Tita P, Pigliaru F, Peraga G, Borretta G, Scaroni C, Bazzoni N, Bianchi A, Berton A, Serban AL, Baldelli R, Fatti LM, Colao A, Arosio M; Italian Study Group of Acromegaly. Acromegaly is associated with increased cancer risk: a survey in Italy. Endocr Relat Cancer. 2017 Sep;24(9):495-504. doi: 10.1530/ERC-16-0553. Epub 2017 Jul 14. PMID 28710115
- [Background] O'Toole SM, Denes J, Robledo M, Stratakis CA, Korbonits M. 15 YEARS OF PARAGANGLIOMA: The association of pituitary adenomas and phaeochromocytomas or paragangliomas. Endocr Relat Cancer. 2015 Aug;22(4):T105-22. doi: 10.1530/ERC-15-0241. Epub 2015 Jun 25. PMID 26113600
- [Background] Beckers A, Aaltonen LA, Daly AF, Karhu A. Familial isolated pituitary adenomas (FIPA) and the pituitary adenoma predisposition due to mutations in the aryl hydrocarbon receptor interacting protein (AIP) gene. Endocr Rev. 2013 Apr;34(2):239-77. doi: 10.1210/er.2012-1013. Epub 2013 Jan 31. PMID 23371967
- [Background] Bilezikian JP, Bandeira L, Khan A, Cusano NE. Hyperparathyroidism. Lancet. 2018 Jan 13;391(10116):168-178. doi: 10.1016/S0140-6736(17)31430-7. Epub 2017 Sep 17. PMID 28923463
- [Result] Jaffrain-Rea ML, Daly AF, Angelini M, Petrossians P, Bours V, Beckers A. Genetic susceptibility in pituitary adenomas: from pathogenesis to clinical implications. Expert Rev Endocrinol Metab. 2011 Mar;6(2):195-214. doi: 10.1586/eem.10.87. PMID 30290451
- [Result] Daly AF, Vanbellinghen JF, Khoo SK, Jaffrain-Rea ML, Naves LA, Guitelman MA, Murat A, Emy P, Gimenez-Roqueplo AP, Tamburrano G, Raverot G, Barlier A, De Herder W, Penfornis A, Ciccarelli E, Estour B, Lecomte P, Gatta B, Chabre O, Sabate MI, Bertagna X, Garcia Basavilbaso N, Stalldecker G, Colao A, Ferolla P, Wemeau JL, Caron P, Sadoul JL, Oneto A, Archambeaud F, Calender A, Sinilnikova O, Montanana CF, Cavagnini F, Hana V, Solano A, Delettieres D, Luccio-Camelo DC, Basso A, Rohmer V, Brue T, Bours V, Teh BT, Beckers A. Aryl hydrocarbon receptor-interacting protein gene mutations in familial isolated pituitary adenomas: analysis in 73 families. J Clin Endocrinol Metab. 2007 May;92(5):1891-6. doi: 10.1210/jc.2006-2513. Epub 2007 Jan 23. PMID 17244780